CLINICAL TRIAL: NCT01872793
Title: Validation of Bioelectrical Impedance Vector Analysis for Nutritional Assessment in Patients With Cirrhosis
Brief Title: Validation of BIVA for Nutritional Assessment in Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, M.D., M.Sc., Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: BIVA02
Record Dates: First submitted 2013-05-24; First posted 2013-06-07 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Liver Cirrhosis; Malnutrition
Keywords: bioelectrical impedance vector analysis; nutritional assessment; nutritional status; mortality; complications
MeSH Terms: conditions — Liver Cirrhosis; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the importance of nutritional status in patient's outcome, there is no gold standard for nutritional assessment. Traditional techniques used in healthy subjects to assess nutritional status cannot be used in cirrhotic patients due especially to ascites and peripheral edema, and altered rates of biochemical markers due to liver failure.

Bioelectrical impedance vector analysis has emerged as a useful method to assess body composition and nutritional status especially in patients at the extremes of body weight (fluid overload, excess of adipose tissue, etc.).

With previous results from our research group, BIVA showed to be useful for evaluating cirrhotic patients.

The aim of this study is to validate our previous results and validate BIVA for nutritional assessment in patients with liver cirrhosis

ELIGIBILITY:
Inclusion Criteria:

Diagnose of liver cirrhosis by two or more of the following criteria:

* Albumin < 3.4 g/dL
* INR ≥ 1.3
* Total bilirubin ≥ 2 mg/dL
* Portal hypertension (esophageal varices, splenomegaly, ascites, etc.)
* Liver biopsy
* Ambulatory patients

Exclusion Criteria:

* Personal history of surgery in the last four weeks
* Thyroid disorders without replacement therapy
* Pregnancy
* Active alcoholism with alcohol ingest in the previous 6 months.
* Acute or chronic renal failure
* Hepatic or renal transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the Gastroenterology Department of a tertiary care setting.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes in nutritional status | At the time of inclusion, every six months up to 36 months
  It will be assessed by bioelectrical impedance vector analysis

OTHER OUTCOMES:
Evaluation of mortality | Through study completion, an average of 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, MD, MSc, Study Chair — Instituto Nacional de Nutrición y Ciencias Médicas "Salvador Zubirán"; Astrid Ruiz-Margain, BSc, MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Ricardo Macías-Rodriguez, MD, MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No